CLINICAL TRIAL: NCT00464724
Title: 3T Perfluorocarbon-Filled Endorectal Magnetic Resonance Spectroscopic Imaging of Prostate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0516; NCI-2011-00517 (Registry Identifier: NCI CTRP); PC061612 (Other: DOD)
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Magnetic Resonance Spectroscopic Imaging; Perfluorocarbon Compound; AIR-MRSI; PFC-MRSI; 3 Tesla; MRSI; PFC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3T MRSI Prostate (Experimental): 3T Magnetic Resonance Spectroscopic Imaging
  Interventions: Procedure: 3T Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Procedure: 3T Magnetic Resonance Spectroscopic Imaging — Part 1 of Study = One MRSI exam with an air-filled endorectal coil (AIR-MRSI) and one with a PFC-filled endorectal coil (PFC-MRSI); Part 2 of Study = MRSI exam with PFC using an endorectal coil only.

SUMMARY:
Objectives:

The objectives of this study are to: 1) evaluate the feasibility of 3T MRSI of prostate in improving the spectral resolution, using a PFC-filled endorectal coil, 2) develop a systematic metabolic grading system for tumor detection by identifying the abnormal peak areas of Cho, Cr, Po, and Ci for the prostate carcinoma, specifically from PFC-filled endorectal 3T MRSI, and 3) evaluate the efficacy of the metabolic grading system in tumor detection.

The long-term goal of the study is to provide an early prognostic indicator and means of monitoring the biologic status of the prostate cancer during the course of the disease.

DETAILED DESCRIPTION:
Part 1:

Prostate cancer tissue has certain differences in its metabolism (chemical makeup) that are not seen in normal tissue. MRSI is a type of magnetic resonance imaging (MRI) that uses the same type of scanner as a standard MRI. Unlike standard MRI, which takes pictures of the body regions, MRSI shows the metabolic features of the prostate cells. MRSI exams that use a "coil" behind the prostate (inside of the rectum) have been used to measure the metabolic features of prostate cancer tissue. This has been shown to improve the accuracy of finding prostate tumor using standard scanners called "1.5T" scanners.

The coil works like an antenna, and air is normally used inside the coil to inflate it. The accuracy of endorectal MRSI exams still needs improvement. Use of PFC instead of air inside of the coil has been shown to greatly improve the quality of MRSI images at 1.5T scanners. At first, researchers want to learn if the newer, stronger (3T) scanners will improve the quality of endorectal MRSI exam when combined with PFC within the coil. PFC is a clear and odorless liquid that, as opposed to air, is physically very similar to human tissue (such as prostate tissue). This makes the MRSI images much clearer.

If you agree to take part in this study (Part 1) and are found to be eligible, you will have 2 MRSI exams (one with air and one with PFC) using an endorectal coil.

Before being inserted, the coil will be inflated with air to check for a possible leak. You will lie on one side, inside of a 3T MRI scanner, and the coil (covered with protective nonlatex or latex) will be inserted into your rectum. Having the coil inserted is similar to having an enema tip inserted. The coil will be filled with air, and you will lie on your back so the first MRSI exam can be completed. Once the first MRSI exam is completed, as much of the air as possible will be removed from the coil using a syringe.

The coil will then be filled with PFC, and the second MRSI exam will be repeated in the same manner. At the end of the exam, the PFC will be removed in the same manner, and then the coil will be removed from the rectum. There will be no direct contact between the PFC or air inside the coil and your body. In total, the 2 MRSI studies should take about 60 minutes.

You will have a prostatectomy (surgical removal of the prostate) within 3 months of having the MRSI exams performed. After the operation, your participation in this study will be over.

Part 2:

Prostate cancer tissue has certain differences in its metabolism (chemical makeup) that are not seen in normal tissue. MRSI is a type of magnetic resonance imaging (MRI) that uses the same type of scanner as a standard MRI. Unlike standard MRI, which takes pictures of the anatomy (body regions), MRSI shows the metabolic features of the prostate. MRSI exams that use a "coil" behind the prostate (inside of the rectum) have been used to measure the metabolic features of prostate cancer tissue. This has been shown to improve the accuracy of prostate tumor detection at standard scanners called "1.5T" scanners.

The coil works like an antenna, and air is normally used inside the coil to inflate it. The accuracy of endorectal MRSI exams still needs improvement. Use of PFC instead of air inside of the coil has been shown to greatly improve the quality of MRSI images at 1.5T scanners. At first, researchers want to learn if the newer, stronger (3T) scanners will improve the quality of endorectal MRSI exam when combined with PFC within the coil. PFC is a clear and odorless liquid that, as opposed to air, is physically very similar to human tissue (such as prostate tissue). This makes the MRSI images much clearer.

If you agree to take part in this study (Part 2) and are found to be eligible, you will have an MRSI exam with PFC using an endorectal coil. Only PFC will be used.

Before being inserted, the coil will be inflated with air to check for a possible leak, and as much as possible of the air will be removed. You will lie on one side, inside of a 3T MRI scanner, and the coil (covered with protective nonlatex or latex) will be inserted into your rectum. Having the coil inserted is similar to having an enema tip inserted. The coil will be filled with PFC, and you will lie on your back so the MRSI exam can be completed. Once the exam is completed, the PFC will be removed from the coil using a syringe and then the coil will be removed from the rectum. There will be no direct contact between the PFC inside the coil and your body. The procedure should take about 30 minutes.

You will have a prostatectomy (surgical removal of the prostate) within 3 months of having the MRSI exam performed. After the operation, your participation in this study will be over.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven, clinical stage 1-3 prostate carcinomas
2. Prostatectomy at M. D. Anderson within 3 months from the time of MRSI
3. An interval of > 6 weeks between the biopsy and MRSI
4. Signed informed consent form

Exclusion Criteria:

1. Contraindications for MRI (e.g. cardiac pacemaker)
2. Contraindications for MRS (e.g. history of abdomino-perineal resection of rectum)
3. Metals or any conditions (e.g. hip prosthesis) that can distort the local magnetic field
4. Previous prostate surgery for prostate carcinoma (including, TURP and cryosurgery), local or systemic treatment for prostate carcinoma (e.g. radiation, androgen deprivation), pelvic radiation (e.g. rectal cancer), rectal surgery, BCG for bladder cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Comparison of linewidths collected from AIR MRSI and PFC-MSRI | 2 MRSI studies should take about 60 minutes; study participation completed with prostatectomy to take place within 3 months of MRSI exams
  The outcome variable for comparing linewidths between the two modalities is paired differences of measurements taken from the same patients. A paired t-test is used to test for a 50% decrease in the mean linewidth as measured by PFC-MRSI versus AIR-MRSI.

CONTACTS AND LOCATIONS:
Overall Officials: Haesun Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org